THE EFFECT OF THERAPEUTIC TOUCH AND MUSIC REST ON SLEEPING APPLIED TO CHILDREN WITH LIVER TRANSPLANTATION

ID: TDK-2020-2358

NCT ID not yet assigned

Initial Release: 09/09/2021

## **Evaluation of Research Data**

Percentage, mean, standard deviation, normal distribution, t-test in independent groups, t-test and ANOVA tests in dependent groups, multiple linear regression and correlation analyzes will be used in the evaluation of the data. Statistical significance level will be accepted as p<0.05.